CLINICAL TRIAL: NCT02408107
Title: Randomised Controlled Trial of a Home-based Physical Activity Intervention in Breast Cancer Survivors
Brief Title: A Home-based Physical Activity Intervention in Breast Cancer Survivors
Acronym: PHAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dudley Group NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ID800
Record Dates: First submitted 2015-03-25; First posted 2015-04-03 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Physical activity; Randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity intervention (Experimental): Received a 30 min physical activity counselling session which employed motivational interviewing to encourage the adoption of current recommended physical activity guidelines. This arm also received 3 support phone calls (1 at the end of months 1, 2 and 3) and a physical activity reminder postcard on months 4 and 5.
  Interventions: Behavioral: Physical activity
- Usual care (No Intervention): This arm received usual care (i.e. no physical activity counselling, support phone calls or post-cards).

INTERVENTIONS:
Behavioral: Physical activity — Physical activity (PA) intervention participants received a 30-45 min face-to-face consultation (1st visit), followed by 15-20 min support telephone calls (end of months 1, 2 and 3). During months 4 and 5 patients received reminder leaflets. Consultations were conducted by the primary researcher after baseline measurements and were based on the four core motivational interviewing principles. The topics covered in the consultation (e.g. goal setting, overcoming barriers, health and safety advice) were similar to other trials that incorporated a PA counselling component. The focus of the follow-up phone calls (end of months 1-3) was to prevent relapse and/or improve maintenance of PA. The intervention participants were encouraged to work towards accumulating at least 30min of moderate-intensity PA on 5-7 days/week.
  Arms: Physical activity intervention

SUMMARY:
The aim of this current study was to investigate the effects of a pragmatic home-based physical activity programme on primarily physical activity levels and secondarily weight maintenance, health-related quality of life (HRQoL), insulin resistance (IR) and lipid concentrations in post-adjuvant therapy breast cancer survivors.

DETAILED DESCRIPTION:
Due to the prevalence of treatment-related health concerns and increased risk of developing metabolic syndrome, recurrence and cardiovascular disease, breast cancer survivors may require diagnostic, therapeutic, supportive or palliative services for many years post-diagnosis. Encouraging breast cancer survivors to adopt a healthy lifestyle post-treatment may reduce the healthcare burden resulting from treatment-related sequelae and improve survival. In particular, higher levels of physical activity (PA) may positively influence some of these side-effects of treatment, enhance quality of life and reduce risk of recurrence and all-cause and breast cancer-related mortality. However, PA levels are generally low among breast cancer survivors and many women decrease their PA following diagnosis. Therefore, interventions are required to improve the post-diagnosis PA levels of breast cancer survivors.

Randomised controlled trials (RCTs) have found improvements in cardiorespiratory fitness, HRQoL, fatigue and weight maintenance in breast cancer survivors participating in PA interventions compared with control groups. However, most of these RCTs utilised facility-based interventions, which may limit their patients who have trouble accessing exercise facilities due to transportation or time-related difficulties. To overcome these problems home-based PA interventions have been investigated and have generally reported good adherence and positive effects on health, fitness and HRQoL outcomes. However, there is a lack of relevant interventions in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 y and over,
* Diagnosed with invasive breast cancer (Stage I-III) within two years of enrolment and no evidence, or clinical suspicion, of metastatic disease,
* Post-surgery and had no surgery planned for the next six months at least,
* Had fully completed adjuvant therapy (radiotherapy and/or chemotherapy) not including hormonal therapy,
* No previous malignancy except in the case of ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), basal cell carcinoma or cervical carcinoma in situ, or where the patient has been disease-free for 10 years,
* No concomitant medical or psychiatric problems that might prevent completion of treatment or follow-up,
* Willing to be randomised, and willing to maintain contact with the investigators over the six months

Exclusion Criteria:

* No evidence of invasive breast cancer (i.e. only pre-invasive disease identified),
* Previous invasive breast cancer (surgically treated DCIS or LCIS is allowed),
* Inability to participate in PA because of severe disability (e.g. severe arthritic conditions), psychiatric illness and vulnerable subjects, such as pregnant women.
* Any other patient where PA was not approved by their oncologist due to the presence of one or more contraindications to exercise in cancer patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Physical activity questionnaire (International Physical Activity Questionnaire) | Baseline and 6 months
  Change in self-reported physical activity (MET-min/wk) from baseline to post-intervention at 6 months in all 80 participants.

SECONDARY OUTCOMES:
Health-related quality of life questionnaire (Functional Assessment of Cancer Therapy (FACT) - Breast) | Baseline and 6 months
  Change in health-related quality of life from baseline to post-intervention at 6 months in all 80 participants.
Body mass | Baseline and 6 months
  Change in body mass (kg) from baseline to post-intervention at 6 months in all 80 participants.
Body Mass Index | Baseline and 6 months
  Change in Body Mass Index (kg/m2) from baseline to post-intervention at 6 months in all 80 participants.
Body fat percentage via bioelectrical impedance analysis | Baseline and 6 months
  Change in body fat percentage (%) from baseline to post-intervention at 6 months in all 80 participants.
Glucose via venepuncture blood samples | Baseline and 6 months
  Change in glucose (mmol/L) assessed using multi-layered slides with the Vitros® 5.1 FS chemistry system from baseline to post-intervention at 6 months in all 80 participants.
Insulin | Baseline and 6 months
  Change in insulin (pmol/L) via a solid phase two-site chemi-luminescence immunometric assay with the Vitros® 5.1 FS chemistry system from baseline to post-intervention at 6 months in all 80 participants.
Insulin Resistance | Baseline and 6 months
  Change in insulin resistance (via Homeostasis Model Assessment) from baseline to post-intervention at 6 months in all 80 participants.
Triglyceride | Baseline and 6 months
  Change in triglycerides (mmol) (via reflectance spectrophotometry) from baseline to post-intervention at 6 months in all 80 participants.
Total cholesterol | Baseline and 6 months
  Change in total cholesterol (mmol) (via reflectance spectrophotometry) from baseline to post-intervention at 6 months in all 80 participants.
High-density lipoprotein cholesterol | Baseline and 6 months
  Change in high-density lipoprotein cholesterol (mmol) (via reflectance spectrophotometry) from baseline to post-intervention at 6 months in all 80 participants.
Low-density lipoprotein cholesterol | Baseline and 6 months
  Change in low-density lipoprotein cholesterol (mmol) (dual chamber package and spectrophotometry) from baseline to post-intervention at 6 months in all 80 participants.
Cardiorespiratory fitness | Baseline and 6 months
  Change in peak oxygen uptake (ml/min/kg) (via gas analysis during exercise tolerance test) from baseline to post-intervention at 6 months in 40% (32) of total recruited.
Systolic blood pressure | Baseline and 6 months
  Change in systolic blood pressure (mmHg) (via automated blood pressure sphygmomanometer) from baseline to post-intervention at 6 months in 40% (32) of total recruited.
Diastolic blood pressure | Baseline and 6 months
  Change in diastolic blood pressure (mmHg) (via automated blood pressure sphygmomanometer) from baseline to post-intervention at 6 months in 40% (32) of total recruited.
Mean Arterial Blood Pressure | Baseline and 6 months
  Change in mean arterial blood pressure (mmHg) (via automated blood pressure sphygmomanometer) from baseline to post-intervention at 6 months in 40% (32) of total recruited.
Resting heart rate | Baseline and 6 months
  Change in resting heart rate (beats/min) (via heart rate telemetry) from baseline to post-intervention at 6 months in 40% (32) of total recruited.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Lahart, PhD, Principal Investigator — University of Wolverhampton; Amtul R Carmichael, MD, Study Director — Russells Hall Hopsital

REFERENCES:
- [Background] Lahart IM, Metsios GS, Nevill AM, Carmichael AR. Physical activity levels in women attending breast screening, receiving chemotherapy and post-breast cancer treatment; a cross-sectional study. Int J Environ Res Public Health. 2014 May 20;11(5):5487-96. doi: 10.3390/ijerph110505487. PMID 24852599
- [Background] Lahart IM, Metsios GS, Nevill AM, Carmichael AR. Physical activity, risk of death and recurrence in breast cancer survivors: A systematic review and meta-analysis of epidemiological studies. Acta Oncol. 2015 May;54(5):635-54. doi: 10.3109/0284186X.2014.998275. Epub 2015 Mar 9. PMID 25752971
- [Background] Rogers LQ, Hopkins-Price P, Vicari S, Pamenter R, Courneya KS, Markwell S, Verhulst S, Hoelzer K, Naritoku C, Jones L, Dunnington G, Lanzotti V, Wynstra J, Shah L, Edson B, Graff A, Lowy M. A randomized trial to increase physical activity in breast cancer survivors. Med Sci Sports Exerc. 2009 Apr;41(4):935-46. doi: 10.1249/MSS.0b013e31818e0e1b. PMID 19276838
- [Background] Payne JK, Held J, Thorpe J, Shaw H. Effect of exercise on biomarkers, fatigue, sleep disturbances, and depressive symptoms in older women with breast cancer receiving hormonal therapy. Oncol Nurs Forum. 2008 Jul;35(4):635-42. doi: 10.1188/08.ONF.635-642. PMID 18591167
- [Background] Pinto BM, Frierson GM, Rabin C, Trunzo JJ, Marcus BH. Home-based physical activity intervention for breast cancer patients. J Clin Oncol. 2005 May 20;23(15):3577-87. doi: 10.1200/JCO.2005.03.080. PMID 15908668
- [Background] Musanti R. A study of exercise modality and physical self-esteem in breast cancer survivors. Med Sci Sports Exerc. 2012 Feb;44(2):352-61. doi: 10.1249/MSS.0b013e31822cb5f2. PMID 21796050
- [Background] Heim ME, v d Malsburg ML, Niklas A. Randomized controlled trial of a structured training program in breast cancer patients with tumor-related chronic fatigue. Onkologie. 2007 Sep;30(8-9):429-34. doi: 10.1159/000104097. Epub 2007 Sep 7. PMID 17848814
- [Background] Vallance JK, Courneya KS, Plotnikoff RC, Yasui Y, Mackey JR. Randomized controlled trial of the effects of print materials and step pedometers on physical activity and quality of life in breast cancer survivors. J Clin Oncol. 2007 Jun 10;25(17):2352-9. doi: 10.1200/JCO.2006.07.9988. PMID 17557948
- [Derived] Lahart IM, Metsios GS, Nevill AM, Kitas GD, Carmichael AR. Randomised controlled trial of a home-based physical activity intervention in breast cancer survivors. BMC Cancer. 2016 Mar 17;16:234. doi: 10.1186/s12885-016-2258-5. PMID 26988367